CLINICAL TRIAL: NCT00593658
Title: Open Label Single Arm Pilot Study of Pentoxifylline in Advanced Hepatopulmonary Syndrome
Brief Title: Pilot Study of Pentoxifylline for Hepatopulmonary Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor tolerability of drug and side effects
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Michael B. Fallon, MD, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F030604005; R03DK065958 (NIH)
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2008-01

CONDITIONS: Hepatopulmonary Syndrome
Keywords: hypoxemia; liver transplantation evaluation; cirrhosis
MeSH Terms: conditions — Hepatopulmonary Syndrome; Hypoxia; Fibrosis | interventions — Pentoxifylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single (Experimental)
  Interventions: Drug: pentoxifylline

INTERVENTIONS:
Drug: pentoxifylline — pentoxifylline extended release 800mg PO TID for 8 weeks

SUMMARY:
The Hepatopulmonary syndrome (HPS) results from intrapulmonary microvascular dilatation that impairs arterial oxygenation in the setting of cirrhosis or portal hypertension. As many as 10-20% of cirrhotics being evaluated for orthotopic liver transplantation (OLT) have advanced HPS and mortality is greater in those with HPS than in those without HPS. Currently, OLT is the only effective treatment, although post-operative mortality in HPS is increased relative to cirrhotic patients without HPS, with a one-year survival of between 68-80 %. Therefore, an effective medical therapy for advanced HPS could improve both pre-operative and post-operative mortality.

Recent work in experimental models of HPS has revealed that both nitric oxide synthase-derived nitric oxide and heme oxygenase-derived carbon monoxide cause intrapulmonary vasodilatation. These alterations appear to be driven in part by TNF-α modulation of pulmonary blood flow and intravascular monocyte accumulation. Pentoxifylline is a nonspecific phosphodiesterase inhibitor with inhibitory effects on TNF-α and has recently been shown to be beneficial in patients with severe alcoholic hepatitis where TNF-α overproduction contributes to liver injury. In experimental HPS, pentoxifylline administration also decreases the severity of oxygenation abnormalities. However, pentoxifylline therapy has been associated with dose limiting side effects in patients with liver disease and the tolerability of pentoxifylline in cirrhotic patients with advanced HPS is unknown. Therefore, this open label single arm clinical trial was designed to evaluate the efficacy and tolerability of 8 weeks of pentoxifylline in cirrhotic patients with advanced HPS being considered for OLT.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing liver transplantation evaluation for cirrhosis
* HPS (positive contrast echocardiography, hypoxemia, no other cause)
* PaO2 < 65mmHg
* ability and willingness to give informed consent

Exclusion Criteria:

* Patients under the age of 19
* active bacterial infections
* known malignancy
* intrinsic cardiopulmonary disease
* known intolerance to pentoxifylline

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-06; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
change in arterial oxygenation (PaO2) and/or alveolar arterial oxygen gradient | 8 weeks

SECONDARY OUTCOMES:
adverse events and safety of pentoxifylline therapy | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Fallon, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Tanikella R, Philips GM, Faulk DK, Kawut SM, Fallon MB. Pilot study of pentoxifylline in hepatopulmonary syndrome. Liver Transpl. 2008 Aug;14(8):1199-203. doi: 10.1002/lt.21482. PMID 18668653